CLINICAL TRIAL: NCT06451445
Title: A Pan-Canadian, Investigator Initiated Clinical Trial With Focal IRE Directed to Intermediate-Risk Prostate Cancer: The WIRED Study
Brief Title: A Pan-Canadian, Investigator Initiated Clinical Trial With Focal IRE Directed to Intermediate-Risk Prostate Cancer
Acronym: WIRED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5926
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IRE Treatment Arm (Experimental): All patients enrolled in this trial will receive IRE treatment with the NanoKnife System.
  Interventions: Device: Irreversible Electroporation (NanoKnife)

INTERVENTIONS:
Device: Irreversible Electroporation (NanoKnife) — Irreversible Electroporation (IRE) using NanoKnife technology uses high voltage current pulses via probes placed around the prostate tumour via the perineum. The electricity damages the cell membranes rendering the cells dead. Hypothesized benefits of IRE over other focal therapy options include the ability to treat large or small lesions. Also, because the technology spares vessels, it can be used to treat prostate areas adjacent to sensitive structures (ie prostate apex near the sphincter and lateral peripheral zone near the neurovascular bundle). Finally, treatments take approximately 1-1.5 hours, thus the technology could be used to treat several patients per day.
  Other Names: NanoKnife System

SUMMARY:
The goal of this clinical trial is to investigate the safety and efficacy of Irreversible Electroporation (IRE) using NanoKnife technology in patients with intermediate-risk prostate cancer. This patient population was chosen because they would otherwise be treated with conventional therapies with high side effects. The main questions it aims to answer are:

1. Is the NanoKnife system is effective at damaging prostate tumour cells, and killing the cancer?
2. Are there any safety concerns with the procedure, or major side effects caused by the treatment?

Participants will undergo IRE treatment with the NanoKnife system, and then complete follow-up appointments for 12-months after the procedure.

DETAILED DESCRIPTION:
Study Population This study is being conducted with intermediate-risk prostate cancer patients (Gleason score 7). This patient population was chosen because they would otherwise be treated with conventional therapies (RP or RT) which are often associated with significant side effects.

Study Design This study is designed to be a prospective, non-randomized study in 100 subjects treated at up to 5 clinical sites in Canada.

Prospective study subjects who sign a written informed consent will be enrolled in the study. Study eligibility will be confirmed at the Screening visit. Transperineal or transrectal prostate biopsy must have been performed no more than 180 days prior to the time of consent. mpMRI must have been within 360 days prior to treatment. If they continue to meet enrollment criteria, they will be scheduled for treatment and after undergoing standard bowel preparation, the NanoKnife System procedure will be carried out under general anesthesia and utilizing transrectal ultrasound (US) guidance.

Subjects will undergo treatment with the NanoKnife System as well as follow-up visits at 1, 3, 6, 9, and 12 months post-procedure. Transrectal US and transperineal or transrectal biopsy will be completed at the 12-month follow up visit. Post-treatment imaging will be completed using mpMRI scan at 9-12 months post-procedure.

Study Agent/ Intervention/ Procedure The intervention being studied is Irreversible Electroporation (IRE) using NanoKnife technology. This technology uses high voltage current via probes placed around the prostate tumour via the perineum. The electricity damages the cell membranes rendering the cells dead. Hypothesized benefits of IRE over other focal therapy options include the ability to treat large or small lesions. Also, because the technology spares vessels, it can be used to treat prostate areas adjacent to sensitive structures (ie. prostate apex near the sphincter and lateral peripheral zone near the neurovascular bundle). Finally, treatments take approximately 1-1.5 hours, thus the technology could be used to treat several patients per day.

Primary Objectives

1. To determine the NanoKnife System's ablation effectiveness and durability by measuring the negative in-field biopsy rate at 12 months.
2. To determine the NanoKnife System's procedural and post-procedural safety profile by evaluating adverse event incidence, type, and severity through 12 months.

Secondary Objectives

1. To evaluate whether clinically significant prostate cancer will develop outside the ablation zone in men selected for focal IRE therapy as determined by positive prostate biopsy outside the ablation zone 12 months post treatment.
2. To evaluate urinary and erectile function after NanoKnife System treatment using validated subject questionnaires (UCLA-EPIC, IPSS, IPSS-QOL, IIEF-15).
3. To determine post-NanoKnife System treatment prostate-specific antigen (PSA) kinetics, including time to PSA nadir and post-nadir PSA stability.
4. To determine the effectiveness of therapy by assessing the need for secondary or salvage treatment following therapy.
5. To determine health-related quality of life (HRQoL) levels after treatment with the NanoKnife System using a validated subject questionnaire (EQ-5D).

Exploratory Objective

1. To evaluate longer term effectiveness of focal IRE and possible delayed adverse events through 5-years.

ELIGIBILITY:
Inclusion Criteria:

1. Is greater than 50 years of age
2. Has at least a 10-year life expectancy
3. Has histologically confirmed organ-confined prostate cancer, clinical stage ≤ T2c
4. Has a PSA ≤ 15 ng/mL or PSA density < 0.15 ng/mL2 if PSA is > 15 ng/mL
5. Has Gleason score 3+4 or 4+3
6. Has no evidence of extraprostatic extension by mpMRI
7. Has no evidence of seminal vesicle invasion by mpMRI
8. Physician is able to visualize prostate gland adequately on transrectal ultrasound imaging during qualifying biopsy
9. Has a transperineal or transrectal targeted prostate biopsy of MRI-visible lesions, plus 10-14 core systematic biopsy confirming Gleason = 7 in MRI target and absence of Gleason ≥ 7 outside target
10. A visible lesion on mpMRI that is accessible to Irreversible Electroporation (IRE) treatment [Note: prostate cancer detected via systematic standard biopsy outside of the adjacent sextant location of the MRI visible lesion will meet entry criterion provided the positive core is Gleason 6; has fewer than 3 prostate biopsy fragments/cores positive]
11. Willing and able to sign a written informed consent form.
12. Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

1. Has known hypersensitivity to pancuronium bromide, atricurium or cisatricurium
2. Is unfit for anesthesia or has a contraindication for agents listed for paralysis
3. Has an active urinary tract infection (UTI)
4. Has a history of bladder neck contracture
5. Is interested in future fertility
6. Has a history (within 3 years) of inflammatory bowel disease
7. Has a concurrent major debilitating illness
8. Had active treatment for a malignancy within 3 years, including malignant melanoma, except for prostate cancer or other types of skin cancer (Note: subjects with untreated active concomitant cancers are excluded, only subjects deemed to be in remission by their cancer care provider for at least three years are eligible)
9. Has any active implanted electronic device (e.g., pacemaker)
10. Is unable or unwilling to catheterize
11. Has had any prior or current prostate cancer therapy, including:

    1. Biologic therapy for prostate cancer
    2. Chemotherapy for prostate cancer
    3. Hormonal therapy for prostate cancer within three months of procedure
    4. Radiotherapy for prostate cancer
    5. Surgery for prostate cancer
12. Has had prior prostate stricture surgery, urethral stent or prostatic implants
13. Has had prior major rectal surgery (except hemorrhoids)
14. Is unfit for pelvic MRI scanning (e.g., severe claustrophobia, permanent cardiac pacemaker, metallic implants that are likely to contribute significant image artifacts, allergy or contraindication to gadolinium (to enhance MRI)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2033-05 (Estimated)

PRIMARY OUTCOMES:
Rate of negative in-field biopsy at 12 months | 1 year
  To determine the NanoKnife System's ablation effectiveness by measuring the negative in-field biopsy rate at 12 months
Incidence of adverse events by type and CTCAE v5.0 severity through 12 months | 1 year
  To determine the NanoKnife System's procedural and post-procedural safety profile by evaluation adverse event incidence, type, and severity through 12 months

SECONDARY OUTCOMES:
Evaluation of clinically significant prostate cancer rate of development outside the ablation zone | 1 year
  To evaluate whether clinically significant prostate cancer will develop outside the ablation zone in men selected for focal IRE therapy as determined by positive prostate biopsy outside the ablation zone 12 months post treatment
Assessment of urinary function after NanoKnife System treatment by comparison of pre- and post-operative UCLA Expanded Prostate Cancer Index Composite | 1 year
  Assessment of urinary function by comparison of pre- and post-operative UCLA Expanded Prostate Cancer Index Composite (UCLA-EPIC) Urinary Domain and International Prostate Symptom Scores (IPSS) and IPSS Quality of Life2 (IPSS-QoL) scores.
Assessment of erectile function after NanoKnife System treatment by comparison of pre- and post-operative IIEF-15 potency scores | 1 year
  Assessment of erectile function by comparison of pre- and post-operative 15-Item International Index of Erectile Function (IIEF-15) potency scores.
Effectiveness of therapy by measurement of prostate-specific antigen (PSA) kinetics | 1 year
  To determine post-NanoKnife System treatment prostate-specific antigen (PSA) kinetics, including time to PSA nadir and post-nadir PSA stability
Assessment of need for secondary or adjuvant treatment | 1 year
  To determine the effectiveness of therapy by collecting data on the number of patients who need secondary or adjuvant treatment within 12-months post-procedure
Evaluation of subject reported pre- and post-operative Quality of Life | 1 year
  To determine health-related quality of life (HRQoL) levels after treatment with the NanoKnife System using a validated subject questionnaire (EQ-5D)

OTHER OUTCOMES:
Evaluation of longer term effectiveness of focal IRE | 5 years
  To examine the rate of progression and re-intervention collected through standard of care follow-up for five years
Collection of data on possible delayed adverse events | 5 years
  To evaluate any delayed adverse events collected through standard of care for five years by type and CTCAE v5.0 severity

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No